CLINICAL TRIAL: NCT00289497
Title: Phase 2 Study for Infrared Thermometry Used by Diabetic Patients at Home
Brief Title: TempTouch IR Thermometry & Diabetic Patient Self-Care
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Diabetica Solutions Inc. (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R44DK054559 (NIH)
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2006-02-09 (Estimated); Status verified 2006-02

CONDITIONS: Diabetic Polyneuropathy; Diabetic Foot Ulcer; Diabetes; Foot Infection
Keywords: Charcot; foot; ulceration; neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetic Foot; Diabetes Mellitus; Ulcer

INTERVENTIONS:
Device: TempTouch®

SUMMARY:
Foot ulcers develop in diabetics with neuropathy because of cumulative injury over the course of several days. These patients do not feel pain, and do not recognize their foot is being injured until a wound develops. Areas about to ulcerate become inflamed and "hot spots" can be identified. This study's purpose is to evaluate the effectiveness of a home infrared temperature probe designed to forewarn patients that an area on the foot is inflamed so they can take preventive measures. The study will evaluate the incidence of diabetic foot ulcers among high-risk patients, evaluate the cost of home temperature monitoring compared to standard therapy, and evaluate patient satisfaction. 180 diabetics at high-risk of having foot complications will be randomized into 3 treatment arms: 1) standard therapy consisting of regular foot care; 2) standard therapy plus recording of a structured foot evaluation using a hand mirror; and 3) standard therapy plus infrared home temperature assessment to identify "hot spots." Device patients will measure temperatures at 6 sites on the foot each day. When temperatures are elevated >4°F patients will contact the research nurse and decrease activity. The primary study outcome will be incident foot ulcers and Charcot fractures.

DETAILED DESCRIPTION:
SIGNIFICANCE & RATIONALE FOR PROPOSED PROJECT Foot problems are the most common complication in diabetics leading to hospitalization.1-5 Approximately one quarter of all hospital days for persons with diabetes are related to foot complications.4,5,8 In the United States there are approximately 120,000 non-traumatic lower extremity amputations performed each year.6,7 In the U.S., 45%-83% of all lower extremity amputations involve diabetics.1,9,5 Overall, patients with diabetes are 15-46 times more likely to have an amputation than patients without diabetes.11,14,15 It has been estimated that 5% to 15% of diabetics will have a lower extremity amputation in their lifetime.11 After their initial amputation 9-17% of diabetic patients will experience a second amputation within the same year12-17 and 25% to 68% of diabetics will have an amputation of the contralateral extremity within five years.18-20 The five-year survival rate after a lower extremity amputation ranges from 41% to 70%.19-21 Indeed, 10% of these patients die before leaving the hospital after a lower extremity amputation.7,9,20 National Initiatives: There are a number of initiatives by federal and state government organizations to prioritize efforts to reduce the burden of diabetes related amputations. Healthy People 2000 and Healthy People 2010 have set a goal of reducing the incidence of diabetes related amputation by 40%, and the U.S. Department of Health and Human Services has prioritized amputation reduction in minorities as one of its strategic Initiatives to Eliminate Racial and Ethnic Disparities in Health. Likewise, the Veterans Administration and Indian Health Service have prioritized amputation prevention for patients with diabetes. For instance, the VA has mandated the development of special programs to evaluate patients with diabetes, identify patients that fit a high-risk profile, and provide specialized treatment programs in order to decrease the impact of diabetes related complications within the Veterans Health Administration. Lower extremity complications in diabetics are common, costly and associated with a high rate of recurrence, morbidity and mortality. Several studies in the U.S. and Europe suggest that amputations and ulcerations can be prevented when special foot care and education are implemented. Despite these types of initiatives, increasing research knowledge, better re-vascularization and diagnostic procedures and an expanding armamentarium of new drugs and technology, the incidence of amputation has increased over the past few decades.15 Precursors to amputation: In diabetes, as in other chronic diseases, patient involvement to identify early warning signs of the disease process is imperative to reduce the incidence of complications and prevent morbidity. Many lower extremity complications involve sensory neuropathy as a pivotal component of the critical pathway for both the development of ulcers and amputations. Therefore, pain and loss of function, primary natural warning systems that alert us to take action and seek medical care, are faulty. Diabetic patients can hence sustain injuries that are not recognized until they are so severe that full thickness ulcerations result. The aim of this study was to further evaluate a tool to help high-risk diabetics identify areas on their feet that are inflamed and prone to ulceration before a wound develops at sites that would otherwise not be recognized as "symptomatic." Results of the Phase I study indicated that high-risk patients with diabetes can effectively use an infrared temperature device to monitor foot temperatures. Patients who used the device had significantly fewer foot complications compared to patients who received education, therapeutic shoes plus insoles and regular foot evaluations alone.

Foot ulcers are one of the most common precursors to diabetes related amputations.8,25 Other factors that have been associated with amputation, such as infection, faulty wound healing, and ischemia, usually do not cause tissue loss or amputation in the absence of a wound. Therefore, ulcer prevention is one of the foci of any amputation prevention program. Three primary pathways or mechanisms of injury have recently been identified in the development of foot ulcers They include wounds that result from ill-fitting shoes (low-pressure injuries that are associated with prolonged or constant pressure from narrow or short shoes), repetitive moderate forces on the sole of the foot, and from puncture wounds (high-pressure injuries with a single exposure of direct pressure). The most common mechanism involves the second scenario (receptive moderate force). Except for puncture wounds, areas that are likely to ulcerate have been associated with increased local skin temperatures due to inflammation and enzymatic autolysis of tissue. Several reports have suggested that wounds develop due to a cumulative effect of unrecognized repetitive injury over the course of several days. Identifying areas of injury by the presence of inflammation would then allow patients or health care providers to take action to decrease the inflammation before a wound develops.

Effectiveness of prevention: Several studies have suggested that foot complications can be prevented by a focused team approach to identify and treat lower extremity complications. This approach generally involves de-weighting pressure areas with special shoes, patient education and self-care practices, re-vascularization, optimal glucose control, infection control, use of appropriate referral patterns, and regular foot care.18, 26-30 Several studies have demonstrated a significant decrease in the incidence of ulceration and re-ulceration when therapeutic footwear, education, and regular diabetic foot care was provided. However, 19-28% of these patients still re-ulcerated within 12-18 months.26,31,32 Edmonds and coworkers18 reported a 26% re-ulceration rate in high-risk diabetics with special shoes and insoles compared to an 83% re-ulceration rate in patients that wore their own shoes. Likewise Uccioli26 reported a 28% re-ulceration rate in diabetics treated with custom shoes and insoles compared to 50% re-ulceration among patients without special footwear. In a descriptive report, Helm and co-workers32 reported a 19% re-ulceration over an 18-month period among patients that healed neuropathic ulcers in total contact casts. As in other studies, after wound closure patients received custom shoes or healing sandals and regular clinical follow-up care. All of these studies were performed at specialty foot centers with a focus on diabetes. Even in these centers, the risk of re-injury was very high.

Predicting impending injury: Our rationale for evaluating skin temperatures involves the search for a quantifiable, reproducible measurement of inflammation that can be used to identify pathologic processes before they result in ulcers. Inflammation is one of the earliest signs of foot ulceration. Five cardinal signs characterize inflammation: redness, pain, swelling, loss of function and heat. Many of these signs are difficult to assess objectively. In the neuropathic extremity, pain and disturbance of function may be absent because of neuropathy and thus are poor indicators of inflammation. In addition, swelling and redness are difficult to objectively grade from clinician to clinician or from visit to visit. Most lay people will not be able to understand or accurately evaluate these subtle parameters. However, temperature measurements can be easily performed by patients or their spouses and provide quantitative information that has been shown to be predictive of impending ulceration in diabetics with sensory neuropathy.

Since ulcers develop as a result of cumulative injury over the course of several days, patients need a mechanism to identify early warning signs of ulceration to prompt them to take appropriate action.44 The high re-ulceration rates reported in previous studies indicate that early warning signs are missed. A home temperature monitoring system for wound prevention is a similar concept to home glucose monitoring to help patients adjust their insulin. In both cases patients need frequent information about a health parameter that has the potential to change in a very short period of time. In both cases patients are taught to use the objective data provided from their home monitoring device to alter their behavior whether it is used to change insulin dosage or activity level. One of the barriers to lowering the incidence of ulcers and amputation is an objective mechanism that patients can use at home, such as a home monitoring system.

In the past, standard patient education focused on teaching patients self-inspection skills that most patients could not adequately perform such as using a hand mirror for visual inspection. In our study of ulcer risk factors, a large proportion of both patients with and without foot ulcers did not have the visual acuity, manual dexterity, or joint flexibility to perform simple self-examination checks of their feet. Among ulcer patients 49% could not position and/or visualize their feet, and 15% of ulcer patients were legally blind in at least one eye. Even if a family member is available to visually inspect the foot, without an objective measure of injury, most laymen will only be able to identify ulcers once they have occurred.33 State of existing knowledge: Over the last three decades, several authors have suggested that skin temperature monitoring may be a valuable tool to detect "at risk" sites in patients who are insensate.34-41 As early as 1971 Goller34 reported an association between increased local temperature and localized pressure leading to tissue injury. Sandrow and coworkers35 subsequently used thermometry as a tool to diagnosis occult neuropathic fractures in patients with diabetes in 1972.

Stess et al.37 and Clark et al.40 described the use of infrared thermography to assess skin temperatures in diabetics, diabetics with neuropathic fractures, diabetics with ulcers, patients with leprosy, and controls. They found that neuropathic foot ulcers frequently had increased skin temperatures surrounding a central necrotic area and suggested that infrared thermometry may be a useful technique to identify patients at risk for ulceration.40 Benbow and coworkers38 took this work a step further and evaluated foot temperatures as a tool to identify diabetics at risk of foot ulceration. They suggested that thermographic patterns could be used to screen high-risk patients.38 They prospectively evaluated 50 patients with diabetes and sensory neuropathy for 3 to 4 years. Six patients developed a neuropathic ulcer during the study period. These patients had significantly higher foot temperatures at baseline than patients who did not ulcerate. All of these early studies used liquid crystal contact thermography to map temperature patterns on the sole of the foot. The devices used in these studies were bulky, expensive and difficult to use or integrate into a normal clinical setting.

In a study at the High-Risk Diabetic Foot Clinic at the University of Texas27 at San Antonio, it was hypothesized that local skin temperatures on the affected limb would be higher in extremities with pathology (neuropathic ulcers, acute Charcot's arthropathy) and the same in patients without pathology when compared to the corresponding site on the contralateral foot. Further, it was expected that temperatures return to normal once ulcer and fracture healing is complete. Lastly, it was questioned whether dermal thermometry could be potentially predictive of neuropathic ulceration. To that end, 143 consecutive patients with diabetes that presented for treatment to the High-Risk Diabetic Foot Clinic were enrolled. All were evaluated with thermometry. These patients were divided into 3 groups: 78 patients with asymptomatic loss of protective threshold, 44 with neuropathic foot ulcerations, and 21 patients with neuropathic (Charcot) fractures. Temperatures were evaluated with a portable handheld infrared skin temperature probe (Dermatemp 1001, Exergen Products, Watertown, MA, USA). Patients' skin temperatures were measured at the time pathology was initially identified and at subsequent clinical follow-up visits for an average of 22.1 ± 6.4 months. Temperatures on the contralateral foot were measured as a control. In this population, there were significant differences in skin temperature in both the Charcot (8.30°F, p < 0.001) and ulcer groups (5.60°F, p < 0.001) compared with the region overlying the site of pathology on the contralateral side. No significant temperature difference was identified in the group with asymptomatic loss of protective threshold group and no acute pathology. Temperatures all normalized at the time of Charcot quiescence and ulcer healing. Eleven percent of patients in the ulcer group re-ulcerated a mean 12.2 ± 6.4 months after initial healing with a corresponding significant increase in skin temperature at the clinic visit immediately preceding reinjury (p < 0.001). These data suggest that monitoring of the corresponding contralateral foot site may provide objective, clinical information before other clinical signs of injury can be identified and that infrared dermal thermometry may be predictive of neuropathic ulceration.27 Subsequent studies have indicated that elevated skin temperatures are directly correlated with location of acute neuropathic osteoarthropathy (Charcot's arthropathy) and that temperatures will equilibrate in a predictable manner as acute Charcot's arthropathy resolves into a quiescent state.28,29 Furthermore, the difference in temperature on the wounded side compared with the corresponding contralateral site decreases as the surface area of the wound decreases.30 As a practical measure, the opposite extremity has been used in previous studies as a control because it is exposed to the same duration and control of diabetes and systemic complications as the affected limb and should represent a built-in comparison source. In this manner, the patient serves as his own control. Because the disease processes of neuropathic fractures and ulceration involves multiple factors that affect lower extremity perfusion and temperature regulation, it would be difficult to identify an absolute skin temperature level that could be considered normal or one that could be used as a universal reference. For instance, the baseline temperatures for a patient with Charcot's fracture may be higher than diabetic patients without this complication or persons without diabetes.45-47 In a related study, temperatures assessed by manual palpation were identified as a relatively inaccurate means of quantifying skin temperature.47 To that end, eleven healthy physicians, eight male with a mean age of 28.6 ± 4.4 years, were enrolled for study. These subjects were instructed to palpate two of five steel cylinders of known temperature using the volar surface of their hands. The five cylinders, arranged randomly were carefully gradated to produce equal, 2, 4 and 6 degree Celsius temperature gradients. They were then asked whether the temperature difference between any two cylinders was equal, 2º, 4º or 6° Celsius. This process was repeated a total of ten times for each participant. Subjects correctly estimated the temperature gradient a mean 1.00 ± 0.89 times out of 10 random attempts. There was not a significant difference between temperature gradient and frequency of correct answers (p > 0.05). It was concluded that, while the laying on of hands in a clinical setting is a necessary and crucial component of the doctor-patient relationship, manual palpation, even in a controlled environment, is not a reliable or objective means to assess temperature.

For this TempTouch IR Thermometry of high-risk diabetic patient self care study the STUDY SPECIFIC AIMS were:

1. To evaluate the effectiveness of a home infrared temperature probe to reduce the incidence of diabetic foot ulcers among high-risk patients;
2. To evaluate the cost of home temperature monitoring compared to standard therapy among high-risk patients with diabetes; and
3. To evaluate patient perceived benefits and satisfaction of home temperature monitoring.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diabetes by WHO criteria
* ability to provide informed consent
* 18-80 years of age

Exclusion Criteria:

* patients with open ulcers or open amputation sites
* active Charcot arthropathy
* severe peripheral vascular disease
* active foot infection
* dementia -impaired cognitive function-
* history of drug or alcohol abuse within one year of the study
* other conditions based on the PI's clinical judgment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2000-06; Study Completion 2003-07

PRIMARY OUTCOMES:
Intervention of device use decreases foot ulcers.

SECONDARY OUTCOMES:
Comparison of foot ulceration from enhanced device group as opposed to control group.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Higgins, DPM, Principal Investigator — Xilas Medical, Inc; C. Mauli Agrawal, Ph.D., Study Director — Xilas Medical, Inc.
Locations (3):
- United States (3):
  - Steven R Beito, DPM, New Braunfels, Texas
  - Robert Wunderlich, DPM, San Antonio, Texas
  - 8800 Village Drive, Suite 202, San Antonio, Texas

REFERENCES:
- [Result] Lavery LA, Higgins KR, Lanctot DR, Constantinides GP, Zamorano RG, Armstrong DG, Athanasiou KA, Agrawal CM. Home monitoring of foot skin temperatures to prevent ulceration. Diabetes Care. 2004 Nov;27(11):2642-7. doi: 10.2337/diacare.27.11.2642. PMID 15504999